CLINICAL TRIAL: NCT01701167
Title: ROMAN (PCA-9000A) PET/CT System Verification
Brief Title: Verification of the Quantitative Accuracy of the PET/CT System Imaging Chain
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Toshiba America Medical Systems, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ROMAN-01
Record Dates: First submitted 2012-10-02; First posted 2012-10-04 (Estimated); Last update posted 2012-10-04 (Estimated); Status verified 2012-10

CONDITIONS: Confirm PCA-9000A PET/CT System is Effective for Its Intended Use

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study will evaluate new technologies that have been included in the new PCA-9000A PET/CT System.

DETAILED DESCRIPTION:
Scope:

To evaluate the new technologies that have been included in the PCA-9000A PET/CT System, the study has the following 3 goals.

* Define and confirm all supported clinical protocols from Low-Dose CT, to PET acquisition and presentation.
* Verification of the quantitative accuracy of the imaging chain.
* Evaluate the performance and stability of the new system and its related quality control and calibration procedures.

Result (Expected):

The study is an essential step in assessing the quality of the hardware and software defining the new PCA-9000A PET/CT System. Several essential parameters for the acquisition, reconstruction, correction, filtering, and presentation will be estimated or adjusted during this period. The evaluation will confirm PCA-9000A PET/CT System is effective for its intended use.

ELIGIBILITY:
Inclusion:

* Patients already scheduled for an FDG test at SDMI
* 40 years and older
* Adult must be able to sign an informed consent form

Exclusion

* Patients not scheduled for an FDG test at SDMI
* 39 years or younger
* Pregnant adult female or plan to be pregnant
* Adult who is unable to sign the informed consent

Min Age: 40 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients already scheduled for a FDG test.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2012-11; Primary Completion 2013-02 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Steinberg Diagnostic Medical Imaging Centers, Henderson, Nevada, United States